CLINICAL TRIAL: NCT03087929
Title: Phase II Follow-up Trial of Rituximab Interferon Transplant Trial: Study Drug-Rituximab and Alpha Interferon
Brief Title: Follow-up Trial of Rituximab Interferon Transplant Trial: Study Drug-Rituximab and Alpha Interferon
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Neil Berinstein, Principal Investigator, Sunnybrook Health Sciences Centre
Other Study IDs: Rituxan INF II
Record Dates: First submitted 2017-02-10; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment Arm: Patients who had previously undergone high dose therapy with stem cell support followed by consolidation with Rituximab and alpha-interferon as part of the trial Treatment of Follicular non-Hodgkin's Lymphoma with High Dose Therapy and Stem Cell Support Followed by Consolidative Immunotherapy with Rituximab and Alpha Interferon. The patients in this arm have consented to long-term follow up.
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up

SUMMARY:
A previous phase II trial entitled Treatment of Follicular non-Hodgkin's Lymphoma with High Dose Therapy and Stem Cell Support Followed by Consolidative Immunotherapy with Rituximab and Alpha Interferon was conducted at the Odette Cancer Centre between 2005 and 2012. The primary objectives of this previous trial was to assess progression free survival and overall survival. Of the 36 patients in this trial, approximately 18 remain in remission. In this new follow up trial, follow up data will prospectively be collected on patients who provide informed consent to do so.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1-2 relapses of WHO Classification follicle centre NHL grade 1-2/3. Patients must have achieved at least a PR to previous treatment.
* Central pathology review before registration
* Ann Arbor stage III or IV
* Measurable disease: defined as clinically or radiologically documented disease with at least one site bidimensionally measurable using clinical exam, CT or MRI performed in the 3 weeks prior to study enrollment.
* ECOG performance status of <2.
* Patients may have received not more than 1 prior course (4 infusions) of rituximab. Timing from last dose of rituximab must exceed 6 months prior to registration. Patients must have demonstrated at least a PR to rituximab if previously administered.
* Patient consent according to institutional and university human experimentation committee requirements
* Adequate Renal, hepatic and hematopoietic function test unless the abnormal values are thought to be due to involvement with lymphoma as defined by:

  * Hb> 85
  * ANC >1000/mm3
  * Platelets >100,000/mm3
  * Serum/Total Bilirubin >=2 SI units
  * AST/ALT <2x Upper Limit of Normal

Exclusion Criteria:

* Positive serology for HIV
* Uncontrolled Infection
* Pregnancy
* CNS Metastases
* History of Psychiatric Disorder
* Other Malignancy (except nonmelanoma skin cancer)
* Serious non-malignant disease (e.g., congestive heart failure, or active uncontrolled bacterial, viral, or fungal infections), or other conditions, which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives.
* Major surgery, other than diagnostic surgery, within four weeks.
* Presence of anti-murine antibody (HAMA) reactivity. These laboratory results must be available prior to receiving treatment for those patients
* who have received prior murine proteins or patients who have allergies to murine proteins.
* New York Heart Association Class III or IV heart disease (see Appendix H, Clinical Evaluation of Functional Capacity of Patients with Heart Disease in Relation to Ordinary Physical Activity) or myocardial infarction within the past six months.
* Treatment with an investigational drug within 30 days or five half-lives (of the study drug with the longest half-life) prior to entry into the study, which ever is longer.
* Previous chemotherapy, immunotherapy, radiotherapy, or investigational therapy for the treatment of other malignancy except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix within the last 5 years.
* History of allergic reactions to compounds chemically related to Rituximab.
* Refusal to practice contraception if of reproductive potential.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twelve patients with low grade follicular lymphoma who consented to long term follow-up and were previously treated with high dose therapy and autologous stem cell transplant with rituximab and alpha interferon as part of the phase II trial Treatment of Follicular Non-Hodgkin's Lymphoma with High Dose Therapy and Stem Cell Support Followed by Consolidative Immunotherapy with Rituximab and Alpha Interferon.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-09-20 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Overall survival | through study completion, up to 15 years
  Number of months from date of enrollment to date of death or last follow-up, whichever comes first.
Progression-free survival | through study completion, up to 15 years
  Number of months from date of enrollment to date of progression. Progression is defined as a greater than or equal to 50% increase in the sum of the product of measurable lesions. Appearance of new lesions will also constitute progressive disease.
Event-free survival | through study completion, up to 15 years
  Number of months from date of enrollment to date of an event. An event is defined as death, disease progression, transformation, or development of secondary malignancy.

SECONDARY OUTCOMES:
Adverse events possibly or probably related to transplant | through study completion, up to 15 years
  Adverse events include second malignancies, myelodysplastic syndrome (MDS), hypogammaglobulinemia, and pulmonary fibrosis. This outcome measurement is descriptive.
Minimal Residual Disease | through study completion, up to 15 years
  This exploratory endpoint is used to evaluate the detection of recurrent lymphoma in peripheral blood DNA. It is measured as real-time quantitative polymerase chain reaction (RQ-PCR) and is expressed as a percent of detection per 100,000 cells at each follow-up time point.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Berinstein, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No